CLINICAL TRIAL: NCT03557515
Title: Reducing Distress in Phase 1 Trial Caregivers: The P1-CaLL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-0514.cc
Record Dates: First submitted 2018-05-22; First posted 2018-06-15 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Caregiver Distress
Keywords: Depression; Cognitive Behavioral Therapy; Coping; Meditation; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Telephonic Sessions (Experimental): All participants will receive four stress management sessions. Then, the participant is randomly assigned to receive 4 weekly additional CBT telephonic sessions. Participants will be given weekly assignments to practice the skills learned in the sessions. Sessions will last 45 minutes to 1 hour. Optional grief and loss telephonic session will be offered.
  Interventions: Behavioral: Stress Management and CBT
- Metta-Meditation Telephonic Sessions (Experimental): All participants will receive four stress management sessions. Then, the participant is randomly assigned to receive 4 weekly additional Metta-meditation sessions. Participants will be given weekly assignments to practice the skills learned in the sessions. Sessions will last 45 minutes to 1 hour. Optional grief and loss telephonic session will be offered.
  Interventions: Behavioral: Stress Management and Metta-Meditation

INTERVENTIONS:
Behavioral: Stress Management and CBT — Stress Management will focus on:
  1. Mind-Body Connection
  2. Coping Skills
  3. Communication
  4. Social Support
  Cognitive Behavioral Therapy will focus on:
  1. Intro to CBT-Tracking Automatic Thoughts
  2. Identifying Distorted Thoughts
  3. Challenging Distorted Thoughts
  4. Core Beliefs/Relapse Prevention
  Arms: CBT Telephonic Sessions
Behavioral: Stress Management and Metta-Meditation — Stress Management will focus on:
  1. Mind-Body Connection
  2. Coping Skills
  3. Communication
  4. Social Support
  Metta-Meditation will focus on:
  1. Intro to Meditation vis Mindfulness of the Breath and Body-Noticing Critical Self Talk
  2. Intro to Brief Loving-Kindness Meditation and Self-Care
  3. Continuing with Additional Metta-Based Exercises to Cultivate Compassion for Oneself and Others and Mitigating Self-Criticism
  4. Review/Plan for Future
  Arms: Metta-Meditation Telephonic Sessions

SUMMARY:
This study seeks to decrease distress in the lives of the caregivers who are helping cancer patients who have entered a phase 1 clinical trial.

DETAILED DESCRIPTION:
This study seeks to decrease distress in the lives of the caregivers who are helping cancer patients who have entered a phase 1 clinical trial. The P1-CaLL study uses a psychosocial intervention aimed at decreasing distress through the utilization of adaptive coping strategies (e.g., meditation, emotion-focused coping) and cognitive behavioral techniques. Caregivers will receive 4 weeks of stress-management sessions (over the phone). Then, they will be randomized to receive 4 more weekly sessions of either Cognitive Behavioral Therapy or Metta-Meditation (over the phone). Participants will receive tasks to complete each week.

ELIGIBILITY:
Inclusion Criteria:

1. Informal caregiver of a patient screening for a phase 1 clinical trial
2. Self-identifies as a caregiver as consistent with the National Study Of Caregiving (NSOC) definition13- individuals who help a patient with self-care, mobility, or household activities (the latter, for health or functioning related reasons) and are either related to the patient (paid or and non-paid) or are unrelated non-paid helpers.
3. Provision to sign and date the consent form.
4. Completes the Patient Health Questionnaire (PHQ-4) screener with a total score of >3.
5. Stated willingness to comply with all study procedures and be available for the duration of the study.
6. Age >18
7. Has consistent access to a telephone
8. Able to read and understand English

Exclusion Criteria:

1. Has a cognitive or psychiatric condition prohibiting participation.
2. Current enrollment in another psychosocial intervention trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Assessing the feasibility of the P1-CaLL intervention by determining the percentage of recruitment and retention | Baseline to end of study period (up to one year)
  Fifty percent of those approached decide to enroll (recruitment), and fifty percent of those enrolled complete all sessions (retention).
Determine the acceptability of the P1-CaLL intervention using a Likert scale | Baseline to end of study period (up to one year)
  Quantitatively measure the acceptability of the P1-CaLL intervention (at least fifty percent of those that complete the intervention rate it) as average or above average on a Likert Scale of Acceptability.

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS) | Baseline to post-assessment (up to 9 weeks)
  The between-subject change in symptoms of distress as measured by response on the Depression Anxiety and Stress Scale (DASS) from baseline (week one) to post-assessment (week nine).
PROMIS-Depression | Baseline to post-assessment (up to 9 weeks)
  Measure between-subject changes in psychosocial variablesin caregivers of phase 1 clinical trial participants.
PROMIS-Anxiety | Baseline to post-assessment (up to 9 weeks)
  Measure between-subject changes in psychosocial variables in caregivers of phase 1 clinical trial participants.
Caregiver Burden (CRA) | Baseline to post-assessment (up to 9 weeks)
  Measure between-subject changes in psychosocial variables in caregivers of phase 1 clinical trial participants.
Positive Benefit Finding (Positive Aspects of Caregiving) | Baseline to post-assessment (up to 9 weeks)
  Measure between-subject changes in psychosocial variables in caregivers of phase 1 clinical trial participants.
Self-Efficacy (CGI) | Baseline to post-assessment (up to 9 weeks)
  Measure between-subject changes in psychosocial variables in caregivers of phase 1 clinical trial participants.
Compassion (Compassion Scale) | Baseline to post-assessment (up to 9 weeks)
  Measure between-subject changes in psychosocial variables in caregivers of phase 1 clinical trial participants.
Dysfunctional Thoughts (ATD) | Baseline to post-assessment (up to 9 weeks)
  Measure between-subject changes in psychosocial variables in caregivers of phase 1 clinical trial participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Kilbourn, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Universtiy of Colorado Denver, Denver, Colorado, United States